

# **Promoting Resilient Youth with Strong Hearts and Minds (PRYSHM)**

Dr. Katie Edwards, Project Leader

Phone. (402) 665-4519 Email. <u>pryshm@unl.edu</u> Website. go.unl.edu/PRYSHM



\*Please allow one business day for us to return calls, texts, emails. If you are in crisis, call 911 OR you can reach out to a 24/7 hotline which are on the resource sheet provided at the end of this survey. You can also get a copy at our website (above).

# TEEN ASSENT/CONSENT FORM

This form tells you more about the research project so that you can decide if you want to be part of it. <u>You</u> **do not** have to get your caregivers' / parents' permission to be part of this project.

# Why are you being asked to be in this research project?

We are asking you to be in this project because you are between the age of 15 and 18 and identify as LGBTQIA2S+ (OR are romantically/sexually interested in people of the same sex/gender as you OR questioning/unsure if you are LGBTQIA2S+).

#### Why are you doing this research project?

LGBTQIA2S+ teens have many strengths and some challenges. We want to make a program for LGBTQIA2S+ teens that help them to use their strengths to overcome things that are hard. Your voice is important in helping us make this program.

#### What are you asking me to do in this research project?

We are asking you to do two things in this project: (1) Take surveys online and (2) Be part of an online program. If you agree to be in this project, we will ask you to take an online survey at three different time points. Each time you take the survey, it will be about 30 minutes. You will do the online program either in between the surveys or after the last survey. This means that some LGBTQIA2S+ teens will get the program pretty soon and other LGBTQIA2S+ teens will get the program in about five months. We use a computer program to randomize who gets the program when, kind of like flipping a coin. You have a 50%

chance of doing the program soon (within a few weeks) or in about five months. You will find out when you will do the program after you take this first survey.

The surveys will ask about things like how you feel about yourself, including your strengths. We will also ask you about your behaviors, like alcohol use, sexual activity, and your relationships, including aggressive behaviors and unwanted sexual experiences.

Before these questions, you will be asked some questions to make sure that you are safe. Because of the nature of the program, we are unable to provide the kind of support that teens who are having strong thoughts or urges to hurt themselves would need. If you are having these experiences, we will reach out to help you get you the kind of support that you need.

The program will have nine sessions, with one session per week, held at the same time every week. There will be options for the program so you can pick the day/time that works best for you. You will learn more about signing up for the program after you take the first survey today if you choose to participate. Each of the nine sessions will be about 60 minutes long. The sessions will happen online on a program called Zoom (we will help you figure out how to work it if you have not used it before). After each of the nine sessions, you will be asked to take a short survey that will take about 5 to 10 minutes. The program sessions are meant to be fun! You will get to meet other LGBTQIA2S+ teens and LGBTQIA2S+ adults (who will teach the classes), do fun activities like watch videos and play games, and learn skills to help you have a healthy and happy future.

So that we can keep track of how well the sessions are going and give feedback to program facilitators, we will video and audio record each session. We will not share these recordings with anyone outside of our research team and will delete the video and audio recordings once we transcribe them into text. We, however, cannot guarantee complete confidentiality because these sessions will be completed as a group. We will emphasize each session that only program participants can attend (no parents, siblings, or friends) and remind teens every session to not share what is said in the group outside of the session.

About halfway through the program, you will be asked to take a brief survey to make sure that you are still doing OK and that you are still safe. The reason we are doing this survey check-in is because unsafe feelings can happen suddenly among some teens. We care about you and other teens and think it is important to make sure that you have not had any changes in these feelings while you are participating in this program. If the check-in survey tells us that you are not safe, we will check in with you. This is the only survey that we will follow up with you about. All of the other surveys that you do we will not follow up with you about, but you can reach out to us if you need help with resources.

Also, we will ask you to give us your contact information when you sign up for this project. If at any point your contact information changes or one of the ways you said was OK to contact you is no longer safe, please reach out to us and we will make sure to update our information so that we only contact you in a way that is OK for you and safe. It is important we be able to contact you to remind you of program sessions and send you the link to the final, online survey.

If you feel safe telling your parent(s) or other people in your life about the project, you can tell them, but you do not have to do so. We will never tell your parents or caregivers or anyone else that you were in the project unless you give us permission to do so. If you are in danger, however, and we contact the police or the trusted adult you tell us, these individuals might tell your parent(s)/caregiver(s) you were in a research project. We will not tell anyone about the nature of the project that you are in. We would



just say that you were participating in a research project. This is because not all LGBTQIA2S+ teens are out, and we care about your safety.

As LGBTQIA2S+ teens participating in this research study, you have certain responsibilities such as (1) coming to the online sessions as scheduled, (2) completing the surveys as requested, and (3) letting us (the research team) know right away if anything negative happens because of being in this research project. Negative things include being upset by anything happening in this project and/or someone like a parent/caregiver finding out that you were in the study, and you getting in trouble or being hurt because of it. We want to know right away if anything like this happens.

### What will you do with the information I tell you?

We will not share what you tell us with other people <u>UNLESS</u> you tell us during a program session or by email/text/phone or in a survey: (1) about a child, including yourself, being hurt or abused, (2) that you plan to hurt yourself or someone else, and/or (3) if someone else, like an elderly or disabled person, is being hurt or abused. If you tell us that you or someone else is in danger, we will have to do a few things to make sure you are safe. Specifically, we will first set up a meeting with you on the phone or on Zoom to get more information about the situation. If after this meeting we are still concerned about someone, including yourself, being hurt or abused, we may then need to contact your trusted adult and/or the authorities (e.g., police, child protective services) in your area about what we know so that they can take the steps to keep people safe. We will tell you that we are doing this, so you know what will happen next.

You should also know that if a parent or another individual in your life contacts us about the project, we will provide them with general information about the project (that it is focused on teaching teens life skills and about healthy choices) and why it is important. We will not provide them with any information about you, including whether you are participating in the study.

Finally, we will share your data, without any information that could identify you, like your name or where you live, in a special database for other scientists who are doing research. Sharing your data helps scientists learn new and important things more quickly than before. Any scientists interested in using your data would have to put in a special request to use it. Any scientist who requests to use your data must promise to keep your data safe and promise not to try to learn your identity. You may decide now or later that you do not want your study data to be added to this database. You can still participate in this research study even if you decide that you do not want your data to be added to the database. If you know now that you do not want your data in the database, please contact us by email or text and let us know. If you decide any time after today that you do not want your data to be added to the database, email or text us, and we will make sure that your study data cannot be shared anymore. Once your data is part of the database, we cannot take back your data that was shared before you changed your mind.

#### How might I feel being in this research project?

Sometimes teens report being sad or feeling awkward when being asked on surveys about their feelings and experiences. Remember that you can skip questions on the surveys that you do not want to answer. After every survey that you take and after each of the program sessions, we will make sure that you know of safe places and people you can contact if you need help for yourself or someone else. You can always reach out to us at any time if you or someone else you know needs help to be safe.

# Do I have to be in this research project?

No, you do not. If you say you do not want to do this project, you will not be in trouble. You can stop being in the project at any time. You can also skip questions that you do not want to answer on the surveys. You



also do not have to talk in the program sessions if you do not want to do so. If you decide you do not want to be in this project anymore, you do not have to tell us why you do not want to be in the project. Deciding not to be in this research study or deciding to withdraw will not affect your relationship with the investigator or with the University of Nebraska-Lincoln. Be aware, that depending on when you withdraw or decide you no longer want to participate, you will only be paid for the surveys you have already completed.

## Will I benefit from being in this research project?

You may not benefit from being in this project. However, some teens tell us that they like to share their ideas and help other people. By being in this project you are helping other LGBTQIA2S+ teens live safe, happy, and healthy lives.

# Will other teens benefit from this research project?

We will ask you questions about what you like about the program and how to make it better for other LGBTQIA2S+ teens. You will also help us make the surveys better. We will take all the feedback that you give us to make the program better before we offer it to LGBTQIA2S+ teens all over the United States! Your voice is so important to us!

### This project has a Certificate of Confidentiality. What does this mean?

To help us protect your privacy while you are in this project, this project has something called a Certificate of Confidentiality from the U.S. Government. We can use this Certificate to legally refuse to provide information that could identify you to others, such as if we received a subpoena (legal document) from a court asking for this information. We would use this Certificate to respond to any orders for information that would identify you, except as explained below: The Certificate cannot be used to refuse a demand for information from people who work for the U.S. Government who want this information to audit (review) projects that receive money or funding from the U.S. Government. You should understand that a Certificate of Confidentiality does not prevent you from providing information to other people about being in this research project. If someone has your written consent (permission) to receive information about your participation in this project, we cannot use the Certificate to refuse to provide that information. We will also still tell state or local authorities (e.g., the police, child protective services) if you tell us about a child (including yourself) being abused or hurt, or if you tell us that you plan to hurt yourself or someone else.

#### What will I get from being in this research project?

We will give you a \$10 gift card for the survey today, a \$20 gift card for the survey you will do in about two months from today, and a \$30 gift card for the survey you will do in about five months from today. You will also get a \$20 gift card for completing a short survey for each program session that you attend. If you opt to receive the gift card through email, you will receive a Visa gift card within a few days. If you opt to receive a gift card through text message, you will receive an Amazon gift card within a few days. If you opt to receive a gift card through mail, you will receive a Visa gift card within a few weeks. In total, you can earn up to \$240 in gift cards for being in this project. Even if you skip survey questions you will still get the gift card. However, you have to get to the end of the survey to get the gift card. You will also still get the gift card if you do not want to talk in the sessions, but you need to stay for the entire session and do the brief survey (you can skip questions) after the session to get the gift card. You also do not have to receive the gift cards if you do not want to do so. You will also get a certificate for completing the program.

IRB# 20220821985FB Date Approved: 09/19/2022 Valid Until: 07/25/2023

# What are my rights as a research subject in this research project?

You may ask any questions about this research project and have those questions answered before agreeing to participate in or during the study. For PRYSHM project related questions, please contact the PRYSHM program office at (402) 665-4519. You can contact us by calling us or texting us. You can also email us if you prefer at <a href="mailto:pryshm@unl.edu">pryshm@unl.edu</a>.

For questions concerning your rights or complaints about the research contact the University of Nebraska - Lincoln Institutional Review Board (IRB): Phone: 1(402)472-6965 Email: <a href="mailto:irb@unl.edu">irb@unl.edu</a>

This study was approved by the University of Nebraska – Lincoln Institutional Review Board.

| Do you want to | be in in this | study? (click one) |
|----------------|---------------|--------------------|
|----------------|---------------|--------------------|

| YES | NO | | | |
|-------------|-----------|---|---|--------------|
| Please type | your name | : | | <br> |
| Date: | | | | _ |
| 37 | C+1 : | C | 1 | <br>/DDVCIII |

You can get a copy of this form on our website at: go.unl.edu/PRYSHM

